CLINICAL TRIAL: NCT02524431
Title: The Changes of Mitochondrial Dynamics and the Molecular Mechanisms in the Trabecular Meshwork of Patients With Glaucoma
Brief Title: The Changes Within the Cells of the Drainage System of the Eye in Patients With Glaucoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain mitochondrial samples
Sponsor: Wills Eye (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, George L. Spaeth MD, Principal investigator, Wills Eye
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-430E
Record Dates: First submitted 2015-08-06; First posted 2015-08-14 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: Mitochondria; trabeculectomy; trabecular meshwork; Glaucoma surgery
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glaucoma subjects (Active Comparator): During glaucoma surgery, collection of trabecular meshwork tissue during surgery that is not needed is cut away from the surgical site. The physician will keep this tissue for analysis by the researchers at Wills Eye Hospital and Thomas Jefferson University Center for Translational Medicine.
  Interventions: Other: Collection of trabecular meshwork tissue during surgery
- Control cadaver eyes (Active Comparator): control cadaver eye are ordered and the collection of trabecular meshwork tissue during surgery and is processed at Thomas Jefferson University
  Interventions: Other: Collection of trabecular meshwork tissue during surgery

INTERVENTIONS:
Other: Collection of trabecular meshwork tissue during surgery — Tissue is collected during surgery at Wills Eye and then processed at thomas jefferson to identify the trabecular meshwork using light microscope. The ocular tissue will be fixed and the mitochondrial cross sections at the longest extent will be measured under electron microscopy (EM) in order to identify the mitochondrial dynamics. Quantitative Polymerase Chain Reaction (qPCR) will be done to identify proteins responsible for mitochondrial fusion.

SUMMARY:
The purpose of this study is to try to identify the cause of damage to the drainage system of the eye (the trabecular meshwork). Damage to this system may cause elevation in the pressure within the eye and thereby damage to the optic nerve and the vision.

DETAILED DESCRIPTION:
During a routine trabeculectomy surgery, a corneo-scleral block that includes TM tissue will be collected at the operating room. This tissue is routinely removed during every trabeculectomy surgery. The tissue will be stored immediately in normal saline at 4 degrees Celsius, and walked directly to the Jefferson Center for Translational Medicine at Thomas Jefferson University by the Wills eye glaucoma research fellow. TM tissue will be identified using light microscope base on TM cell pigmentation. The ocular tissue will be fixed and placed in pre-cooled fixative on ice for 1 hour. The lengths of mitochondrial cross sections at the longest extent will be measured under electron microscopy (EM) in order to identify the mitochondrial dynamics. Quantitative Polymerase Chain Reaction (qPCR) will be done to identify proteins responsible for mitochondrial fusion.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 2-year diagnosis of POAG
* Moderate to advanced stage of the disease
* DDLS stages 5 through 10 with visual field loss
* Age between 21 and 80 years
* Planned trabeculectomy with or without concomitant cataract surgery

Exclusion Criteria:

* Age ≤ 20 years old
* Any other type of glaucoma other than POAG
* Patients who had undergone selective laser trabeculoplasty (SLT) or argon laser trabeculoplasty (ALT)
* Patients with history of ocular trauma
* Patients with previous eye surgery will be excluded both from the study and the control groups

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
3-D EM tomography for mitochondria obtained from sample tissue | 1 year

SECONDARY OUTCOMES:
Gene expression of Drp1 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George Spaeth, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes